CLINICAL TRIAL: NCT00928954
Title: Investigation and Treatment of Ocular Motor Disorders: Cross-over Comparison of Gabapentin and Memantine as Treatment for Nystagmus
Brief Title: Cross-over Comparison of Gabapentin and Memantine as Treatment for Acquired Nystagmus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, John Leigh, R. John Leigh, M.D., Case Western Reserve University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NIHR01EY06717; NIHR01EY06717 (Other: National Eye Institute); NIH R01 EYO6717 (Other Grant/Funding Number: National Eye Institute)
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Nystagmus
Keywords: gabapentin; memantine; nystagmus; Drug treatment
MeSH Terms: conditions — Nystagmus, Pathologic | interventions — Gabapentin; Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin (Active Comparator): Increasing dose to 300 mg four times per day (total of 1200 mg/day)
  Interventions: Drug: gabapentin
- Memantine (Active Comparator): Increasing dose over two weeks to 20 mg twice/day (total of 40 mg/day).
  Interventions: Drug: memantine

INTERVENTIONS:
Drug: gabapentin — increasing to 1200 mg/day
  Other Names: Neurontin
  Arms: Gabapentin
Drug: memantine — increasing to 40 mg/day
  Other Names: Nameda
  Arms: Memantine

SUMMARY:
Involuntary oscillations of the eyes (nystagmus) impairs vision so that affected patients, who have neurological disorders such as Multiple Sclerosis (MS) , cannot read or watch TV. Two medicines have been reported to suppress nystagmus and improve vision in such patients: gabapentin and memantine. The investigators set out to test which of these two drug was more effective by carrying out a double-blind cross-over study. In this way, we could determine which drug worked best in each patient.

DETAILED DESCRIPTION:
The study entails careful measurements of visual acuity and precise measurements of eye movements, using a contact lens device (magnetic search coil method). In this way, it is possible to make objective and reliable measurements of the effect of each drug, which are unbiased by the investigator or the patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older) males or females with acquired nystagmus that is degrading their vision

Exclusion Criteria:

* Pregnant women
* Individuals who cannot describe their visual symptoms, cooperate with testing, or give informed consent
* Individuals with intolerance of gabapentin or memantine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Leigh, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- Veterans Affairs Medical Center, 10701 East Boulevard, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin First and Then Memantine; Memantine First, Then Gabapentin: Increasing dose to 300 mg four times per day (total of 1200 mg/day) for the gabapentin.
  Increasing dose over two weeks to 20 mg twice/day (total of 40 mg/day) for memantine.
Period: Overall Study
Arm/Group | Gabapentin First and Then Memantine | Memantine First, Then Gabapentin
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Increasing dose to 300 mg four times per day (total of 1200 mg/day) for the gabapentin.
  Increasing dose over two weeks to 20 mg twice/day (total of 40 mg/day) for memantine.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in logMAR Visual Acuity of Each Eye, Measured During Far or Near Viewing
Time Frame: After 2 weeks of therapy, for both drugs
Measure: Number; unit: logMAR
Arm/Group | Gabapentin | Memantine
Number analyzed (Participants) | 10 | 10
logMAR
  Participant 1, Right Eye | 0 | 0.1
  Participant 1, Left Eye | 0.2 | 0.2
  Participant 2, Right Eye | 0.1 | 0.2
  Participant 2, Left Eye | 0.2 | 0
  Participant 3, RIght Eye | -0.1 | -0.2
  Participant 3, Left Eye | NA — Below level of detection | NA — Below level of detection
  Patricipant 4, RIght Eye | 0.3 | -0.1
  Participant 4, Left Eye | 0.1 | 0.1
  Participant 5, Right Eye | 0.1 | 0.2
  Particpant 5, Left Eye | 0 | 0.1
  Particpant 6, RIght Eye | 0.4 | 0
  Particpant 6, Left Eye | 0.2 | 0.2
  Particpant 7, Right Eye | -0.1 | 0.1
  Particpant 7, Left Eye | 0.1 | 0.1
  Participant 8, Right Eye | 0.1 | 0
  Participant 8, Left Eye | 0 | 0.1
  Particpant 9, Right Eye | 0 | 0
  Participant 9, Left Eye | 0 | 0
  Participant 10, Right Eye | -0.1 | 0.3
  Participant 10. Left Eye | 0.1 | 0.2

2. Primary Outcome: Percent Change in Median Eye Speed
Description: Median eye speed during attempted visual fixation by each eye
Time Frame: After 2 weeks of therapy, for both drugs
Measure: Number; unit: Percent change
Arm/Group | Gabapentin | Memantine
Number analyzed (Participants) | 10 | 10
Percent change
  Participant 1, Right Eye | -59.1 | -21.5
  Participant 1, Left Eye | -69.8 | -35.1
  Participant 2, Right Eye | -19.9 | -26.0
  Participant 2, Left Eye | -19.8 | -35.5
  Participant 3, RIght Eye | -53.5 | -44.6
  Participant 3, Left Eye | -41.3 | -40.2
  Patricipant 4, RIght Eye | -72.8 | -8.6
  Participant 4, Left Eye | -76.6 | 11.4
  Participant 5, Right Eye | -56.6 | -35.5
  Particpant 5, Left Eye | -42.0 | -26.5
  Particpant 6, RIght Eye | -26.0 | -44.8
  Particpant 6, Left Eye | -25.9 | -29.5
  Particpant 7, Right Eye | 49.5 | -29.0
  Particpant 7, Left Eye | 26.5 | -24.1
  Participant 8, Right Eye | -0.9 | -60.4
  Participant 8, Left Eye | -0.7 | -24.8
  Particpant 9, Right Eye | -39.5 | 2.2
  Participant 9, Left Eye | -44.1 | -19.4
  Participant 10, Right Eye | 159 | -80.6
  Participant 10. Left Eye | 104.4 | -79.3

ADVERSE EVENTS:
Arm/Group | Gabapentin | Memantine
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes